CLINICAL TRIAL: NCT04862299
Title: Pelvic-perineal Disorders in Women With Sphincter Tears, a Retrospective Study
Brief Title: Pelvic-perineal Disorders in Women With Sphincter Tears
Acronym: PAPOASI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PAPOASI
Record Dates: First submitted 2021-04-15; First posted 2021-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Obstetrical Perineal Injury and Anal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to INSEE, in 2016, in France, there were 785,000 births. According to the latest national perinatal survey in 2016, 80.4% of women gave birth by vaginal delivery. Of these, 52.1% had perineal tears and 0.8% had 3rd and 4th degree tears. Of these 3rd and 4th degree tears, 2.2% occurred during instrumental delivery and 0.5% during spontaneous delivery. In recent years, there has been an increase in the prevalence of obstetric anal sphincter injuries. Mc Pherson et al. found a prevalence of LOSA (Obstetric Anal Sphincter Injury) of 2% in 2004 versus 4.6% in 2008. Gurol-Urganci et al. also found an increase in prevalence from 1.8% in 2000 to 5.9% in 2012. This increase is probably due to improved diagnosis by obstetrical teams. Indeed, a large number of LOSAs remained undiagnosed at birth and these occult lesions were subsequently found by endoanal ultrasound. In the Andrews et al. study, when women were reexamined, the prevalence of LOSA increased from 11% to 24.5%. As practitioner training improved, the prevalence of LOSA at birth became increasingly accurate. Obstetric anal sphincter injuries are responsible for significant physical and psychological morbidity. These obstetrical lesions of the anal sphincter can generate functional consequences (including anal incontinence in the first rank), which will have harmful effects on the quality of life of the women, they can involve a social isolation passing by the limitation of displacements and physical and social activities. The daily life of these women can remain impacted by the consequences of LOSA until more than 10 years after delivery. In addition, a loss of self-esteem as well as feelings of guilt, shame and frustration are reported in these women. Thus, some will speak of a LOSA syndrome, which includes emotional, social and psychological consequences, including the ability to assume one's role as a mother. LOSA are perineal tears corresponding to the 3rd and 4th degree, formerly and respectively called complete perineum and complicated complete perineum. The Sultan classification for perineal tears proposed in 1999 was adopted by the Royal College of Obstretricians and Gynecologists (RCOG) and is the most widely used in the scientific literature worldwide. It defines the 3rd degree as a perineal injury involving the anal sphincter complex alone.

Anal continence is a balance between several factors such as rectal sensitivity, stool quality, the smooth and striated muscles of the anal sphincter, the pubo-rectal muscle webbing and the innervation of these structures. Obstetrical trauma of the stretching and compression type affects all these structures. All of these lesions can contribute to the development of anal incontinence. However, these structures are not routinely evaluated in women who have had an obstetric anal sphincter injury.

Pelvic-perineal pain was studied in 2 studies and involved 24.7% to 35% of women with obstetric anal sphincter injuries.

Compared to women without LOSA, women with LOSA had a later return to sexual intercourse, with more severe anal incontinence during the first week after LOSA. Indeed, at 12 weeks postpartum, the rate of women who resumed sexual intercourse was lower in the group of women with LOSA than in the group without LOSA.

The pelvic-perineal disorders faced by women with LOSA affect their quality of life, their sexuality, and their health. Thus, early identification of all pelvic-perineal disorders appears to be a priority in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with an obstetric anal sphincter injury diagnosed in the delivery room
* Patients referred for a pre-rehabilitation perineal assessment between June 2016 and February 2021
* French-speaking patient

Exclusion Criteria:

* Patient with occult obstetric anal sphincter injury
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of her data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient whose age is ≥ 18 years, with an obstetric anal sphincter injury diagnosed in the delivery room, referred for a pre-rehabilitation perineal assessment between June 2016 and February 2021
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Clinical pictures of pelvic-perineal disorders in women | Year 1
  This outcome corresponds to the symptoms presented by the patient (Urinary Symptoms scores: Urinary Symptom Profil Score (USP, It consists of 13 items that assess stress urinary incontinence, urge urinary incontinence, and obstructive symptoms.), anal incontinence: St Marks Score, St Mark's Incontinence score for assessment of anal incontinence following obstetric anal sphincter injuries (OASIS), Score 0-4: minimal, score 5-12: moderate, 13-19: severe, >20: major).

SECONDARY OUTCOMES:
Prevalence of these lesions | Year 1
  This outcome corresponds to the number of sphincter injuries found in the delivery room.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie BILLECOQ, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Groupe Hospitalier Paris Saint-Joseph, France

REFERENCES:
- [Background] McPherson KC, Beggs AD, Sultan AH, Thakar R. Can the risk of obstetric anal sphincter injuries (OASIs) be predicted using a risk-scoring system? BMC Res Notes. 2014 Jul 24;7:471. doi: 10.1186/1756-0500-7-471. PMID 25056485
- [Background] Gurol-Urganci I, Cromwell DA, Edozien LC, Mahmood TA, Adams EJ, Richmond DH, Templeton A, van der Meulen JH. Third- and fourth-degree perineal tears among primiparous women in England between 2000 and 2012: time trends and risk factors. BJOG. 2013 Nov;120(12):1516-25. doi: 10.1111/1471-0528.12363. Epub 2013 Jul 3. PMID 23834484
- [Background] Andrews V, Sultan AH, Thakar R, Jones PW. Occult anal sphincter injuries--myth or reality? BJOG. 2006 Feb;113(2):195-200. doi: 10.1111/j.1471-0528.2006.00799.x. PMID 16411998
- [Background] Cornell K, De Souza A, Tacey M, Long DM, Veerasingham M. The effect of implementing a new guideline and operative pro forma on the detection and management of third- and fourth-degree perineal tears. Int J Womens Health. 2016 May 5;8:131-5. doi: 10.2147/IJWH.S101188. eCollection 2016. PMID 27226734
- See also: Related Info — https://www.em-consulte.com/article/1253328/definitions-epidemiologie-et-facteurs-de-risque-de